CLINICAL TRIAL: NCT02484586
Title: Dispensing Study to Assess the Visual Performance of Optimised Prototype Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRTC2014-04
Record Dates: First submitted 2015-06-24; First posted 2015-06-29 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Presbyopia; Refractive Error
Keywords: Presbyopia; Refractive error; Contact lens
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Presbyope group (Other): 40 years and over with a reading add.
  Control lens: Etafilcon A, Nelfilcon A, Nesofilcon A, Somofilcon A, 58% Poly-HEMA
  Test lens: Etafilcon A
  Up to 10 prototype contact lens designs and at least 1 commercially available contact lens designs will be worn by each participant for up to a week on a daily disposable modality. Participants will attend separate fitting and assessment visits for each lens type (Fitting Visit on Day 1, and Assessment Visit as late as Day 7, but may be as early as 6 hours after the Fitting Visit). There will be a minimum 1 night washout period between lens designs, i.e. after an assessment visit but before the next fitting visit.
  Interventions: Device: Etafilcon A; Device: Nelfilcon A; Device: Nesofilcon A; Device: Somofilcon A; Device: 58% Poly-HEMA
- Non-Presbyope group (Other): 18-39 years with no reading add.
  Control lens: Etafilcon A, Nelfilcon A, Omafilcon A
  Test lens: Etafilcon A
  Up to 10 prototype contact lens designs and at least 1 commercially available contact lens designs will be worn by participants for up to a week on a daily disposable modality. Participants will attend separate fitting and assessment visits for each lens type (Fitting Visit on Day 1, and Assessment Visit as late as Day 7, but may be as early as 6 hours after the Fitting Visit). There will be a minimum 1 night washout period between lens designs, i.e. after an assessment visit but before the next fitting visit.
  Interventions: Device: Etafilcon A; Device: Nelfilcon A; Device: Omafilcon A

INTERVENTIONS:
Device: Etafilcon A — Prototype lens material
Device: Etafilcon A — Control lens for presbyope group
  Other Names: 1-Day Acuvue Moist Multifocal
  Arms: Presbyope group
Device: Nelfilcon A — Control lens for presbyope group
  Other Names: Dailies Aqua Comfort Plus Multifocal
  Arms: Presbyope group
Device: Nesofilcon A — Control lens for presbyope group
  Other Names: Biotrue ONEday for Presbyopia
  Arms: Presbyope group
Device: Nelfilcon A — Control lens for non-presbyope group
  Other Names: Dailies Aqua Comfort Plus
  Arms: Non-Presbyope group
Device: Etafilcon A — Control lens for non-presbyope group
  Other Names: 1-Day Acuvue Moist
  Arms: Non-Presbyope group
Device: Somofilcon A — Control lens for presbyope group
  Other Names: Clariti 1 Day Multifocal
  Arms: Presbyope group
Device: 58% Poly-HEMA — Control lens for presbyope group
  Other Names: SEED 1dayPure moisture Multistage
  Arms: Presbyope group
Device: Omafilcon A — Control lens for non-presbyope group
  Other Names: Proclear Multifocal
  Arms: Non-Presbyope group

SUMMARY:
The aim of this study is to assess the visual performance of multiple optimised prototype soft contact lens designs compared to commercially available contact lenses.

DETAILED DESCRIPTION:
Prospective, double-masked, crossover, bilateral wear, dispensing clinical trial where participants will wear multiple prototype (test) and commercial (control) lenses.

Multiple prototype contact lens designs will be assessed against commercial control lenses during the study, where each design will be worn for up to a week. There will be a minimum 1 night washout period between lens designs.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent.
* Be at least 18 years old, male or female.
* Willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator.
* Have ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses.
* Is correctable to at least 6/12 (20/40) or better in each eye with contact lenses.
* Be suitable and willing to wear contact lenses.

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition (including infection or disease) of the cornea, conjunctiva or eyelids that would preclude contact lens fitting and safe wearing of contact lenses.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjogrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment. Ocular medication can be prescribed during the course of the trial as per standard optometric practice.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial. Note: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.
* Eye surgery within 12 weeks immediately prior to enrolment for this trial.
* Previous corneal refractive surgery.
* Contraindications to contact lens wear.
* Known allergy or intolerance to ingredients in any of the clinical trial products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity on a LogMAR (logarithm of the minimum angle of resolution) scale | Approximately 1 week after lens fitting
  For each lens, visual acuity will be measured at distance with a computerised LogMAR chart and at near with a near LogMAR chart. Data will be summarised as means +/- standard deviations. No transformation is likely to be required. Visual acuity will be compared between each lens design and control lens types. The significance of lens design will be determined for each visit.
  Repeated effects linear mixed model with subject random intercepts or paired t tests will be employed for the analysis of visual acuity. Analysis will be performed within each study arm namely presbyopes and non-presbyopes.

SECONDARY OUTCOMES:
Subjective rating of vision on a 1-10 visual analogue scale | Approximately 1 week after lens fitting
  For each lens, subjective ratings of vision will be assessed with a questionnaire based on a 1 to 10 scale in steps of 1. The questionnaire has been designed specifically for this study. Data will be summarised as means +/- standard deviations. No transformation is likely to be required. Subjective ratings will be compared between each lens design and control lens types. The significance of lens design will be determined for each visit. Repeated effects linear mixed model with subject random intercepts or paired t tests will be employed for the analysis of subjective ratings. Analysis will be performed within each study arm namely presbyopes and non-presbyopes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sha, BOptom/BSc, Principal Investigator — Brien Holden Vision Institute
Locations (1):
- Brien Holden Vision Institute, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Jong M, Tilia D, Sha J, Diec J, Thomas V, Bakaraju RC. The Relationship between Visual Acuity, Subjective Vision, and Willingness to Purchase Simultaneous-image Contact Lenses. Optom Vis Sci. 2019 Apr;96(4):283-290. doi: 10.1097/OPX.0000000000001359. PMID 30907859
- [Derived] Sha J, Tilia D, Kho D, Amrizal H, Diec J, Yeotikar N, Jong M, Thomas V, Bakaraju RC. Visual Performance of Daily-disposable Multifocal Soft Contact Lenses: A Randomized, Double-blind Clinical Trial. Optom Vis Sci. 2018 Dec;95(12):1096-1104. doi: 10.1097/OPX.0000000000001311. PMID 30451806